CLINICAL TRIAL: NCT01903239
Title: Long Term Prospective Study Evaluating Effectiveness of Narrow Margins for Low-Risk Head and Neck Basal Cell Carcinomas
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Thomas Jefferson University (Other)
Collaborators: Advanced Aesthetics (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB#11D.479
Record Dates: First submitted 2013-02-15; First posted 2013-07-19 (Estimated); Last update posted 2016-02-05 (Estimated); Status verified 2016-02

CONDITIONS: Basal Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Basal Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Low-Risk BCC Excisional Margins (Other): This is a study investigating the efficiency of 1-2 mm margins for the excision of low-risk basal cell carcinoma.
  Interventions: Procedure: Low-Risk BCC Excisional Margins

INTERVENTIONS:
Procedure: Low-Risk BCC Excisional Margins — After the head and neck basal cell carcinomas satisfy the National Comprehensive clinical and histopathological criteria, all tumors are excised at the 2 mm margin.

SUMMARY:
The purpose of this study is to determine the narrowest excision margin for head and neck Basal Cell Carcinoma (BCC) tumors satisfying the National Comprehensive Cancer Network® (NCCN) low-risk for recurrence clinical and histopathological criteria that gives an acceptable (95%) clinical cure-rate over a 3 year follow-up period. Margins of 1 and 2mm are evaluated.

DETAILED DESCRIPTION:
Basal Cell Carcinoma (BCC) is the most common skin cancer in the US. Most are treated by surgical excision. Excision margins vary by tumor size, anatomic location, histological subtype, and surgeon preference. Published recommendations and follow up observation times vary. Current clinical practice supports the 4 mm excision margin; however, this can be a disservice to the patient by potentially excising additional normal tissue unnecessarily and yielding larger scars. Considering healthcare costs, both the excision and repair components are usually billed by size measurements. Determining the narrowest excision margin to give an acceptable clinical cure could feasibly reduce this expenditure.

ELIGIBILITY:
Inclusion Criteria:

* Patient has a BCC <10mm on their cheeks, forehead, scalp & neck or <6mm on their central face, eyelids, eyebrows, periorbital, nose, lips, chin, mandible, preauricular & postauricular, temple & ear
* The BCC has well defined borders
* The BCC is primary
* The Patient is not immunosuppressed
* The BCC is not located at a site of prior radiation therapy
* The histologic subtype is nodular or superficial
* There is no perineural involvement

Exclusion Criteria:

* Patient has a BCC >or=10mm on their cheeks, forehead, scalp & neck or >or=6mm on their central face, eyelids, eyebrows, periorbital, nose, lips, chin, mandible, preauricular & postauricular, temple & ear
* The BCC has poorly defined borders
* The BCC is recurrent
* The Patient is immunosuppressed
* The BCC is located at a site of prior radiation therapy
* The histologic subtype is aggressive
* There is perineural involvement

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 179 (Estimated)
Dates: Start 2011-11; Primary Completion 2017-01 (Estimated); Study Completion 2017-01 (Estimated)

PRIMARY OUTCOMES:
Success rate of narrow (1 and 2mm)margin excision of low-risk facial BCC | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Jason B Lee, MD, Principal Investigator — Jefferson Dermatology Associates
Locations (2):
- United States (2):
  - Advanced Aesthetics, Bensalem, Pennsylvania
  - Jefferson Dermatology Associates, Philadelphia, Pennsylvania